CLINICAL TRIAL: NCT07227441
Title: Chronic Infections and Inflammation in ME/CFS: An Observational Study
Acronym: CHIIME
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 24-43260
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Keywords: ME/CFS; myalgic encephalomyelitis; chronic fatigue syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, peripheral blood mononuclear cells, plasma, serum, nasal swab, stool, and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-COVID ME/CFS: Individuals who received a diagnosis of ME/CFS prior to the beginning of SARS-CoV-2 pandemic and whom SARS-CoV-2 was not expected to be the driver of ME/CFS
- Post-COVID ME/CFS: Individuals who received a diagnosis of ME/CFS following the beginning of the SARS-CoV-2 pandemic and in who SARS-CoV-2 was expected to be the driver of ME/CFS
- Healthy control: Individuals who have overlapping demographic characteristics (age, sex, race, and other factors determined by PI) with participants who have ME/CFS

SUMMARY:
CHIIME is a study of people who have myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS). People who do not have this condition will also be enrolled. Volunteers will be observed and sampled over time to identify the long-terms biological drivers and impact of their condition. The overall goal is to understand the biological and physiological mechanisms that are driving this condition.

DETAILED DESCRIPTION:
CHIIME is an observational, prospective study of individuals who have myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS). The overall objective of the study is to investigate the clinical characteristics and biological signatures of ME/CFS over time by performing deep clinical phenotyping with high-quality biospecimen collection and curation of individuals with and without the condition.

Enrolled volunteers will be seen at San Francisco General Hospital. Visits include a detailed interview, biospecimen collection, and various assessments. No personal identifiers are used for specimen bank samples.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* At least 18 years of age
* Either: (1) a reported diagnosis of ME/CFS or (2) no history of ME/CFS or other infection-associated chronic conditions (healthy control)

Exclusion Criteria:

* Self reported or documented chronic anemia with hemoglobin <9 g/dL
* Known HIV, hepatitis B, or hepatitis C infection
* Diagnosis of an infection-associated chronic condition other than ME/CFS or Long COVID (e.g. chronic Lyme disease, post-Ebola syndrome, etc.)
* Serious medical or psychiatric illness that, in the opinion of the site investigator, would interfere with the ability to adhere to study requirements or to give informed consent
* Active drug or alcohol use or dependence that, in the opinion of the PI, would interfere with adherence to study requirements or to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll individuals with a diagnosis of ME/CFS across a wide spectrum of age, race, gender, and disease severity and will also enroll a subset of people without ME/CFS or other infection associated chronic conditions (healthy control)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Participant Sex | Baseline Visit
  The proportion of men and women participating in the baseline visit.
Participant Age | Baseline Visit
  The median age of study participants at enrollment.
Participant race/ethnicity | Baseline Visit
  The proportion of participants from each demographic group.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Peluso, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No